CLINICAL TRIAL: NCT02522780
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Investigating the Efficacy and Safety of Mesalamine 2 g Extended Release Granules (Sachet) for Maintenance of Clinical and Endoscopic Remission in Ulcerative Colitis
Brief Title: Mesalamine 2 g Sachet for the Maintenance of Clinical and Endoscopic Remission in Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000175; 2015-002558-11 (EudraCT Number)
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2019-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalamine (Experimental): Mesalamine 2 g extended release granules (sachet), administered orally once daily (QD) for 6 months.
  Interventions: Drug: Mesalamine
- Placebo (Placebo Comparator): Placebo matched to mesalamine extended release granules (sachet), administered orally QD for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine — Pharmaceutical form: Granules in sachet; Route of administration: Oral use
  Other Names: Mesalazine; Pentasa
  Arms: Mesalamine
Drug: Placebo — Pharmaceutical form: Granules in sachet; Route of administration: Oral use
  Arms: Placebo

SUMMARY:
The purpose of this trial was to investigate the safety and efficacy of mesalamine 2 g extended release granules (sachet) once a day (QD) for maintenance of clinical and endoscopic remission in subjects with UC. The duration of treatment for each subject was 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years, with Ulcerative Colitis in remission

Exclusion Criteria:

* Evidence of other forms of inflammatory bowel disease
* Infectious disease (including human immunodeficiency virus [HIV], hepatitis B virus [HBV], or hepatitis C virus [HCV])
* Disease limited to proctitis <15 cm
* Short bowel syndrome
* Prior colon resection surgery
* History of severe/fulminant UC
* Intolerant or allergic to aspirin or salicylate derivatives
* Use of rectal formulations (5-aminosalicylic acid [5-ASA], steroids) within ≤7 days
* Women who are pregnant or nursing
* History of known malignancy
* History of bleeding disorders, active gastric or active duodenal ulcers, autoimmune diseases, or mental/ emotional disorders, that would interfere with their participation in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (96):
- United States (18):
  - Preferred Research Partners, Little Rock, Arkansas
  - United Research Institute, Murrieta, California
  - Research Associates of South Florida, LLC, Miami, Florida
  - IMIC, Palmetto Bay, Florida
  - Medical Research Center of Florida, Pembroke Pines, Florida
  - Lenus Research and Medical Group, Sweetwater, Florida
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Associates in Gastroenterology, PLC, Hermitage, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - BI Research Center, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - DM Clinical Research, Tomball, Texas
  - Advanced Research Institute, Ogden, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Digestive & Liver Disease Specialists, Norfolk, Virginia
- Bulgaria (9):
  - Multiprofile Hospital For Active Treatment Avis Medica, Pleven
  - University Multiprofile Hospital for Active Treatment Kaspela, Plovdiv
  - Medical Center Excelsior OOD, Sevlievo
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
  - Medical Center Asklepion - Humane Medicine Research EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Diagnostic Consultative Centre Mladost M OOD, Varna
- Canada (2):
  - Topstone Research Institute, Ottawa, Ontario
  - Toronto Digestive Disease Associates Inc, Toronto, Vaughan
- Hungary (7):
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Semmelweis Egyetem Institute, Budapest
  - Vasútegészségügyi Nonprofit Kiemelten Közhasznú Kft. Debreceni Egészségügyi Központja, Debrecen
  - ENDOMEDIX Kft., Miskolc
  - Karolina Korhaz Rendelointezet, Mosonmagyaróvár
  - Clinfan Kft., Szekszárd
- Latvia (5):
  - Polana-D, LTD, Daugavpils
  - Digestive Diseases Centre Gastro, Riga
  - Latvian Maritime Medicine Centre, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Mexico (3):
  - ICARO Investigaciones en Medicina, S.A de C.V, Chihuahua City
  - Maria Auxiliadora Hospital, Guadalajara
  - Investigación Biomédica para el Desarrollo de Fármacos, S.A. de C.V., Zapopan
- Poland (12):
  - Osrodek Medycyny Rodzinnej Sp. z o.o., Sobótka, Lower Silesian Voivodeship
  - Lexmedica, Wroclaw, Lower Silesian Voivodeship
  - Zespół Przychodni Specjalistycznych PRIMA Sp. z o.o., Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Intermed, Częstochowa
  - Economicus - NZOZ ALL-MEDICUS, Katowice
  - Investigational site, Ksawerów
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lodz
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Endoskopia Sp. z o.o., Sopot
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Russia (14):
  - Regional Clinical Hospital, Krasnoyarsk
  - City Clinical Hospital # 51, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - Research Institute of Physiology of Sibirian Branch the RAMS, Novosibirsk
  - Omsk State Medical Academy, Omsk
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan Regional Clinical Hospital, Ryazan
  - State Budget Institution of Ryazan region" Regional Clinical Hospital", Ryazan
  - City Hospital #31, Saint Petersburg
  - City Polyclinic #38, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Medical Company "Hepatolog", LLC, Samara
  - Stavropol State Medical Academy, Stavropol
- Serbia (3):
  - Clinical Hospital Centar Zvezdara, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Health Center Valjevo, Valjevo
- Switzerland (3):
  - Inselspital Bern, Bern
  - Investigational site, Bern
  - Universitätsspital Zürich, Zurich
- Ukraine (20):
  - Kyiv Municipal Clinical Hospital #18, Kyiv, Kyïv
  - Medical Center LLC Ukrainian German Antiulcer Gastroenterology Center BIK Kyiv, Kyiv, Kyïv
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Municipal Institution Dnipropetrovsk Regional Clinical Hospital n.a. I.I. Mechnykov, Dnipropetrovsk
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #2, Kharkiv
  - SI National Institute of Therapy n.a. L.T. Mala of National Academy of Medical Sciences of Ukraine, Kharkiv
  - Municipal Intitution "Kherson City Clinical Hospital n.a. A. and O. Tropinykh", Kherson
  - Private Enterprise Private Manufactire Company "Acinus", Kirovohrad
  - Kremenchuk city Hospital # n.a O.T.Bohaievskyi, Kremenchuk
  - Kyiv City Clinical Hospital #8, Kyiv
  - Kyiv Municipal Clinical Hospital #18, Kyiv
  - Medical Center Universal Clinic Oberih of LLC Kapytal, Kyiv
  - Municipal City Clinical emergency Hospital, Lviv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
  - Small Business Private Enterprise Medical Center "Pulse", Vinnytsia
  - Vinnytsia Regional Clinical Hospital Hospital n.a. M.I. Pyrohov, Vinnytsia
  - Municipal Institution 6th City Clinical Hospital of Zaporizhzhia City Council, Zaporizhzhia
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhia
  - Medical Centre of PE First Private Clinic, Zhytomyr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 sites in 10 countries randomized subjects to this trial between February 2016 to April 2018, the last subject completed last visit in September 2018. Of 403 subjects screened, 276 subjects were randomized in a 1:1 ratio to either mesalamine or placebo group (138 subjects each), for 6 months.
Pre-assignment Details: Of 276 subjects, (a) 53 were rolled-over from Trial 000174 (NCT02522767) who achieved remission after 8-weeks double-blind treatment with placebo (Pathway 1a; 4 subjects) or mesalamine (Pathway 1b; 10 subjects), or an additional 8-weeks open-label treatment with mesalamine (Pathway 2; 39 subjects), and (b) 223 subjects were de novo (Pathway 3).
Period: Overall Study
Arm/Group | Mesalamine | Placebo
Started | 138 | 138
Treated | 137 | 135
Intention-to-treat (ITT) Population | 136 | 136
Completed | 121 | 111
Not Completed | 17 | 27
Not completed — Consent withdrawn by subject | 5 | 7
Not completed — Protocol deviation | 1 | 3
Not completed — Subject refused endoscopic procedure | 0 | 1
Not completed — Adverse event, non-fatal | 11 | 16

BASELINE CHARACTERISTICS:
Population: The ITT analysis set included all randomized subjects who were assigned to mesalamine 4 g extended release granules in Trial 000174 (NCT02522767) (Pathway 1b) or randomized via Pathways 2 or 3.
Groups:
- Mesalamine: Mesalamine 2 g extended release granules (sachet), administered orally QD for 6 months.
- Total: Total of all reporting groups
Arm/Group | Mesalamine | Placebo | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 130 | 126 | 256
  >=65 years | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (13.50) | 45.2 (13.65) | 43.4 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 77 | 147
  Male | 66 | 59 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 130 | 127 | 257
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 130 | 130 | 260
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.56 (4.812) | 24.89 (4.657) | 24.73 (4.729)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Remission at Month 6
Description: The proportion of subjects with remission was defined by Clinical and Endoscopic Response Score: 0 for rectal bleeding; 0 or 1 for stool frequency; 0 or 1 for endoscopic score. The Clinical and Endoscopic Response Score ranged between 0 (normal) to 9 (severe disease), higher scores indicating greater disease severity. The score included clinical response component to assess subject's symptoms and endoscopic response component to assess objective evidence of inflammation. Clinical response component had two subscales: stool frequency ranging from 0 (normal number of stools) to 3 (>=5 stools more than normal) and rectal bleeding ranging from 0 (no blood seen) to 3 (blood alone passes). The Endoscopic response component had one subscale: flexible sigmoidoscopy/colonoscopy ranging from 0 (normal) to 3 (severe disease). Data is presented cumulative for all pathways.
Time Frame: Month 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo.
Number analyzed (Participants) | 136 | 136
Participants | 82 | 67
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Proportions were compared between treatment groups at Month 6; Test type: Superiority; p > 0.05, Cochran-Mantel-Haenszel — The p-value was based on Cochran-Mantel-Haenszel test by controlling pathway of randomization, at a 0.05 significance level; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.96 to 2.54]

2. Secondary Outcome: Proportion of Subjects in Clinical Remission at Month 2, 4, and 6
Description: The proportion of subjects in clinical remission was defined as a score of 0 for rectal bleeding and 0 or 1 for stool frequency based on clinical response score component of the Clinical and Endoscopic Response Score. Clinical response score component had two subscales to assess subject's symptoms: rectal bleeding ranging from 0 (no blood seen) to 3 (blood alone passes) and stool frequency ranging from 0 (normal number of stools) to 3 (>=5 stools more than normal). The scores of clinical response component ranged from 0 (normal) to 6 (severe disease), higher scores indicating greater disease severity. Data is presented cumulative for all pathways.
Time Frame: Month 2, 4, and 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 136 | 136
Participants
  Month 2 | 122 | 116
  Month 4 | 113 | 113
  Month 6 | 96 | 89
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Proportions were compared between treatment groups over 6 months; Test type: Superiority; p > 0.05, Generalised estimating equation approach — The p-value was based on Generalized estimating equations (GEE) approach with binary outcomes (clinical remission) and an unstructured working correlation matrix, at a 0.05 significance level; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.76 to 2.03]

3. Secondary Outcome: Time to Relapse
Description: Time to relapse was defined as the number of days from randomization to the day of withdrawal due to escalation of therapy. Data is presented cumulative for all pathways.
Time Frame: Time from randomization to the day of withdrawal due to escalation of therapy (up to 6 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 136 | 136
days | NA [NA to NA] — Median and 95% confidence interval (CI) was not estimable due to insufficient events to meet the threshold for 50% on the Kaplan-Meier curve. | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient events to meet the threshold for 50% on the Kaplan-Meier curve.
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Times to relapse were compared between treatment groups up to 6 months; Test type: Superiority; p > 0.05, Log Rank — The p-value was based on log-rank test using pathway of randomization as the stratification factor, at a 0.05 significance level; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.25 to 1.44]

4. Secondary Outcome: Proportion of Subjects With an Increase From Baseline in the Clinical and Endoscopic Response Score by 2 or More Points in at Least 1 Component or by 1 or More Points in at Least 2 Components at Month 6
Description: The proportion of subjects with an increase from baseline in the Clinical and Endoscopic Response Score by 2 or more points in at least 1 component, or by 1 or more points in at least 2 components were reported. The Clinical and Endoscopic Response Score ranged between 0 (normal) to 9 (severe disease), higher scores indicating greater disease severity. The score included clinical response component to assess subject's symptoms and endoscopic response component to assess objective evidence of inflammation. Clinical Response component had two subscales: stool frequency ranging from 0 (normal number of stools) to 3 (>=5 stools more than normal) and rectal bleeding ranging from 0 (no blood seen) to 3 (blood alone passes). The Endoscopic Response component had one subscale: flexible sigmoidoscopy/colonoscopy ranging from 0 (normal) to 3 (severe disease). Data is presented cumulative for all pathways.
Time Frame: Month 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 136 | 136
Participants | 14 | 30
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Proportions were compared between treatment groups at Month 6; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.19 to 0.79]

5. Secondary Outcome: Change From Baseline in Serum C-reactive Protein (CRP) Levels at Month 2, 4, and 6
Description: The adjusted mean change from baseline in serum CRP levels at Month 2, 4, and 6 were reported. Data is presented cumulative for all pathways.
Time Frame: Baseline, Month 2, 4, and 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 136 | 136
mg/L
  Month 2: number analyzed (Participants) | 127 | 121
  Month 2 | 0.8 (4.76) | 2.2 (15.63)
  Month 4: number analyzed (Participants) | 123 | 113
  Month 4 | 1.0 (5.69) | 0.9 (5.53)
  Month 6: number analyzed (Participants) | 116 | 106
  Month 6 | 0.8 (3.67) | 2.5 (16.66)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Adjusted mean treatment difference in CRP levels over 6 months was reported; Test type: Superiority; p > 0.05, ANCOVA — The p-value was based on a repeated-measures analysis of covariance (ANCOVA) model with an unstructured correlation matrix , at a 0.05 significance level; Mean difference = -1.0, 95% CI 2-sided [-2.7 to 0.7]

6. Secondary Outcome: Change From Baseline in Fecal Calprotectin Levels at Month 2, 4, and 6
Description: The adjusted mean change from baseline in fecal calprotectin levels at Month 2, 4, and 6 were reported. Data is presented cumulative for all pathways.
Time Frame: Baseline, Month 2, 4, and 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mcg/g
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 136 | 136
mcg/g
  Month 2: number analyzed (Participants) | 127 | 118
  Month 2 | -94.8 (553.00) | 12.8 (509.70)
  Month 4: number analyzed (Participants) | 121 | 113
  Month 4 | -41.7 (533.02) | 53.6 (581.64)
  Month 6: number analyzed (Participants) | 114 | 103
  Month 6 | -43.5 (553.13) | 36.4 (559.98)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Adjusted mean treatment difference in fecal calprotectin levels over 6 months was reported; Test type: Superiority; p > 0.05, ANCOVA — The p-value was based on a repeated-measures ANCOVA model with an unstructured correlation matrix, at a 0.05 significance level; Mean difference = -66.92, 95% CI 2-sided [-140.2 to 6.36]

7. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Scores at Months 2, 4, and 6
Description: The IBDQ is an instrument used to assess quality of life in adult subjects with ulcerative colitis. It includes 32 questions on 4 domains of Health-Related Quality-of-Life (HRQOL): Bowel Systems (10 items), Emotional Function (12 items), Social Function (5 items), and Systemic Function (5 items). Subjects were asked to recall symptoms and quality of life from the last 2 weeks and rate each item on a 7-point Likert scale (1=worst to 7=best). The total IBDQ was computed as the sum of the responses to the individual IBDQ questions. The total score can range between 32 to 224 with higher scores indicating a better HRQOL. The adjusted mean change from baseline at Month 2, 4, and 6 for the IBDQ total scores were reported. Data is presented cumulative for all pathways.
Time Frame: Baseline, Month 2, 4, and 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: points on a score
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 136 | 136
points on a score
  Month 2: number analyzed (Participants) | 113 | 116
  Month 2 | -1.3 (17.78) | -0.4 (20.00)
  Month 4: number analyzed (Participants) | 114 | 111
  Month 4 | -0.6 (20.40) | -0.3 (18.53)
  Month 6: number analyzed (Participants) | 105 | 101
  Month 6 | -0.5 (24.80) | -1.2 (23.44)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Adjusted mean treatment difference in IBDQ total scores over 6 months was reported; Test type: Superiority; p > 0.05, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean difference = -0.32, 95% CI 2-sided [-4.41 to 3.77]

8. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a subject participating in a clinical trial. Any AEs includes serious as well as non-serious AEs. An SAE is defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect, or was an important medical event. Any AE which occurred in the time interval from initial dosing (investigational medicinal product [IMP] intake) to the end of treatment visit (Month 6) was considered treatment-emergent. Data is presented cumulative for all pathways.
Time Frame: Up to Month 6
Population: The analysis was based on safety analysis set which included all subjects who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 137 | 135
Participants
  Any Treatment-Emergent AEs | 42 | 49
  Treatment-Emergent SAEs | 2 | 3

9. Secondary Outcome: Severity of Adverse Events
Description: The number of subjects with intensity of AEs (classified as mild, moderate or severe) were presented. Data is presented cumulative for all pathways.
Time Frame: Up to Month 6
Population: The analysis was based on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 137 | 135
Participants
  Mild | 32 | 32
  Moderate | 18 | 22
  Severe | 2 | 3

10. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Laboratory Values: Hematology
Description: Proportion of subjects with markedly abnormal changes from baseline in hematology values are presented. Criteria for markedly abnormal laboratory (Hematology): Basophils/Leukocytes: >=5%, Eosinophils/Leukocytes: >=10%, Erythrocytes: <=3.5*10^6/μL, Hematocrit: <=0.32%; >=0.56%, Hemoglobin: <=11.5 g/dL, Leukocytes: <=2.8*10^3/μL; >=16.0*10^3/μL, Lymphocytes/Leukocytes: <=10%; >=80%, Monocytes/Leukocytes: >=20%, Neutrophils/Leukocytes: <=15%; >=90%, Platelets: <=75*10^3/μL; >=700*10^3/μL. Data is presented cumulative for all pathways.
Time Frame: Baseline, Month 6
Population: The analysis was based on safety analysis set. Here, 'Number Analyzed' signifies number of subjects with available data at specified category for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 137 | 135
Participants
  Basophils/Leukocytes: >=5%: number analyzed (Participants) | 135 | 135
  Basophils/Leukocytes: >=5% | 0 | 1
  Eosinophils/Leukocytes: >=10%: number analyzed (Participants) | 135 | 135
  Eosinophils/Leukocytes: >=10% | 3 | 7
  Erythrocytes: <=3.5*10^6/μL: number analyzed (Participants) | 135 | 135
  Erythrocytes: <=3.5*10^6/μL | 2 | 1
  Hematocrit: <=0.32%: number analyzed (Participants) | 135 | 135
  Hematocrit: <=0.32% | 1 | 0
  Hematocrit: >=0.56%: number analyzed (Participants) | 135 | 135
  Hematocrit: >=0.56% | 8 | 12
  Hemoglobin: <=11.5 g/dL: number analyzed (Participants) | 135 | 135
  Hemoglobin: <=11.5 g/dL | 29 | 23
  Leukocytes: <=2.8*10^3/μL: number analyzed (Participants) | 135 | 135
  Leukocytes: <=2.8*10^3/μL | 4 | 4
  Leukocytes: >=16.0*10^3/μL: number analyzed (Participants) | 135 | 135
  Leukocytes: >=16.0*10^3/μL | 2 | 0
  Lymphocytes/Leukocytes: <=10%: number analyzed (Participants) | 135 | 135
  Lymphocytes/Leukocytes: <=10% | 3 | 4
  Lymphocytes/Leukocytes: >=80%: number analyzed (Participants) | 135 | 135
  Lymphocytes/Leukocytes: >=80% | 0 | 0
  Monocytes/Leukocytes: >=20%: number analyzed (Participants) | 135 | 135
  Monocytes/Leukocytes: >=20% | 0 | 1
  Neutrophils/Leukocytes: <=15%: number analyzed (Participants) | 135 | 135
  Neutrophils/Leukocytes: <=15% | 0 | 0
  Neutrophils/Leukocytes: >=90%: number analyzed (Participants) | 135 | 135
  Neutrophils/Leukocytes: >=90% | 0 | 0
  Platelets: <=75*10^3/μL: number analyzed (Participants) | 135 | 134
  Platelets: <=75*10^3/μL | 0 | 0
  Platelets: >=700*10^3/μL: number analyzed (Participants) | 135 | 134
  Platelets: >=700*10^3/μL | 1 | 0

11. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Laboratory Values: Coagulation
Description: Proportion of subjects with markedly abnormal changes from baseline in coagulation values are presented. Criteria for markedly abnormal laboratory (coagulation): Activated Partial Thromboplastin Time (aPTT): >70 seconds (sec), Prothrombin International Normalized Ratio (INR): <0.8; >1.1. Data is presented cumulative for all pathways.
Time Frame: Baseline, Month 6
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 137 | 135
Participants
  aPTT: >70 sec: number analyzed (Participants) | 133 | 131
  aPTT: >70 sec | 0 | 0
  Prothrombin INR: <0.8: number analyzed (Participants) | 133 | 130
  Prothrombin INR: <0.8 | 0 | 2
  Prothrombin INR: >1.1: number analyzed (Participants) | 133 | 130
  Prothrombin INR: >1.1 | 46 | 54

12. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Laboratory Values: Serum Chemistry
Description: Proportion of subjects with markedly abnormal changes from baseline in serum chemistry values are presented. Criteria for markedly abnormal laboratory (serum chemistry): Alanine Aminotransferase (ALT): >3*upper limit of normal (ULN), Alkaline Phosphatase (ALP): >3*ULN and 25% increase (inc) from baseline (BL), Aspartate Aminotransferase (AST): >3* ULN, Bilirubin: >=1.5* ULN, Blood Urea Nitrogen: >=10.7 mg/dL, Calcium: <=1.8 mg/dL; >=3.9 mg/dL, Chloride: <=90 mmol/L; >=115 mmol/L, Creatinine: >=177 mg/dL, Gamma Glutamyl Transferase: >3*ULN, Glomerular Filtration Rate (GFR): <30 mL/min, Glucose: <=2.8 mg/dL; >=10 mg/dL, Potassium: <=3.0 mmol/L; >=5.8 mmol/L, Sodium: <=130 mmol/L; >=155 mmol/L. Data is presented cumulative for all pathways.
Time Frame: Baseline, Month 6
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 137 | 135
Participants
  ALT: >3*ULN: number analyzed (Participants) | 135 | 135
  ALT: >3*ULN | 1 | 1
  ALP: >3*ULN & 25% inc from BL: number analyzed (Participants) | 135 | 135
  ALP: >3*ULN & 25% inc from BL | 0 | 0
  AST: >3*ULN: number analyzed (Participants) | 135 | 135
  AST: >3*ULN | 2 | 2
  Bilirubin: >=1.5*ULN: number analyzed (Participants) | 135 | 135
  Bilirubin: >=1.5*ULN | 8 | 5
  Blood Urea Nitrogen: >=10.7 mg/dL: number analyzed (Participants) | 135 | 135
  Blood Urea Nitrogen: >=10.7 mg/dL | 8 | 11
  Calcium: <=1.8 mg/dL: number analyzed (Participants) | 135 | 135
  Calcium: <=1.8 mg/dL | 0 | 0
  Calcium: >=3.9 mg/dL: number analyzed (Participants) | 135 | 135
  Calcium: >=3.9 mg/dL | 9 | 12
  Chloride: <=90 mmol/L: number analyzed (Participants) | 135 | 135
  Chloride: <=90 mmol/L | 0 | 0
  Chloride: >=115 mmol/L: number analyzed (Participants) | 135 | 135
  Chloride: >=115 mmol/L | 0 | 0
  Creatinine: >=177 mg/dL: number analyzed (Participants) | 135 | 135
  Creatinine: >=177 mg/dL | 0 | 0
  Gamma Glutamyl Transferase: >3*ULN: number analyzed (Participants) | 135 | 135
  Gamma Glutamyl Transferase: >3*ULN | 6 | 4
  GFR: <30 mL/min: number analyzed (Participants) | 111 | 109
  GFR: <30 mL/min | 0 | 0
  Glucose: <=2.8 mg/dL: number analyzed (Participants) | 135 | 135
  Glucose: <=2.8 mg/dL | 0 | 0
  Glucose: >=10 mg/dL: number analyzed (Participants) | 135 | 135
  Glucose: >=10 mg/dL | 11 | 14
  Potassium: <=3.0 mmol/L: number analyzed (Participants) | 135 | 135
  Potassium: <=3.0 mmol/L | 0 | 0
  Potassium: >=5.8 mmol/L: number analyzed (Participants) | 135 | 135
  Potassium: >=5.8 mmol/L | 0 | 2
  Sodium: <=130 mmol/L: number analyzed (Participants) | 135 | 135
  Sodium: <=130 mmol/L | 0 | 0
  Sodium: >=155 mmol/L: number analyzed (Participants) | 135 | 135
  Sodium: >=155 mmol/L | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Month 6
Description: Treatment-Emergent AEs were defined as AEs which occurred in the time interval from initial dosing (IMP intake) to the end of treatment visit.
Arm/Group | Mesalamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/135
Serious Adverse Events (participants affected / at risk) | 2/137 | 3/135
Other Adverse Events (participants affected / at risk) | 23/137 | 28/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesalamine (N=137) | Placebo (N=135)
Hypertension (Vascular disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Ecthyma (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mesalamine (N=137) | Placebo (N=135)
Glomerular filtration rate decreased (Investigations) | 1 | 5
Alanine aminotransferase increased (Investigations) | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 1
Faecal calprotectin increased (Investigations) | 3 | 1
Colitis ulcerative (Gastrointestinal disorders) | 14 | 20
Respiratory tract infection viral (Infections and infestations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT02522780/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT02522780/SAP_001.pdf